CLINICAL TRIAL: NCT01341470
Title: A Single- and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2495655 in Japanese Subjects
Brief Title: A Study of LY2495655 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 14270; I1Q-JE-JDDH (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — landogrozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Single IV dose LY2495655 (Experimental): Single 70 milligram (mg) dose LY2495655 administered intravenously (IV)
  Interventions: Drug: LY2495655
- Multiple SC dose 17.5 mg LY2495655 (Experimental): 17.5 mg of LY2495655 administered subcutaneously (SC) every 2 weeks for 8 weeks (total of 5 doses)
  Interventions: Drug: LY2495655
- Multiple SC dose 140 mg LY2495655 (Experimental): 140 mg of LY2495655 administered subcutaneously (SC) every 2 weeks for 8 weeks (total 5 doses)
  Interventions: Drug: LY2495655
- Multiple SC dose 420 mg LY2495655 (Experimental): 420 mg dose of LY2495655 administered subcutaneously (SC) every 2 weeks for 8 weeks (total 5 doses)
  Interventions: Drug: LY2495655
- Single IV dose placebo (Placebo Comparator): Single Placebo dose administered intravenously (IV)
  Interventions: Drug: Placebo
- Multiple SC dose placebo (Placebo Comparator): Placebo dose administered subcutaneously (SC) every 2 weeks for 8 weeks (total of 5 doses)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY2495655 — administered intravenously or subcutaneously
  Arms: Multiple SC dose 140 mg LY2495655; Multiple SC dose 17.5 mg LY2495655; Multiple SC dose 420 mg LY2495655; Single IV dose LY2495655
Drug: Placebo — administered intravenously or subcutaneously
  Arms: Multiple SC dose placebo; Single IV dose placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple doses of LY2495655 administered subcutaneously and intravenously in Japanese subjects.

ELIGIBILITY:
Inclusion Criteria

* Single dose cohort

  * Overtly healthy males or females, as determined by medical history and physical examination
  * Between the ages of 24 and 50 years
* Multiple dose cohorts

  * Sedentary males and females with stable medical problems, if any, that, in the investigator's opinion, will not place the subject at increased risk by participating in the study and will not interfere with interpretation of the data
  * Between the ages of 50 and 85 years
  * Score <600 Metabolic Equivalent Tasks (METs) per week based on International Physical Activity Questionnaire (IPAQ)
* All subjects

  * Male subjects: agree to use a reliable method of birth control
  * Female subjects: women not of child-bearing potential due to surgical sterilization (at least 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history, or menopause
  * Up to third generation Japanese, that is defined as all of the subject's biological grandparents are of exclusive Japanese descent and have been born in Japan
  * Are ambulatory and able to perform a stair climb test
  * Have clinical laboratory tests within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
  * Have venous access sufficient to allow for blood sampling and/or administration of investigational product for intravenous administration

Exclusion Criteria:

* Single dose cohort

  * Intend to use over the counter or prescription medication within 14 days prior to dosing through 2 months after dosing except for thyroid replacement hormones or non-absorbed topical preparations per investigator instructions
  * Abnormal supine blood pressure defined as diastolic blood pressure > 90 millimeters of mercury (mmHg) and/or systolic blood pressure >140 mmHg
* Multiple dose cohort

  * If taking medications, subjects who have not been stable for at least 3 months, or the time required to produce stable effects of the drug
  * Abnormal supine blood pressure defined as >100 mmHg and/or systolic blood pressure >160 mmHg
* All subjects

  * Have known allergies to LY2495655, related compounds or any components of the formulation
  * Have a history or presence of cardiovascular, respiratory (including moderate to severe restrictive lung disease and obstructive disease, chronic bronchitis, and those with symptomatic asthma), hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of constituting a risk when taking the study medication or of interfering with the interpretation of data
  * Have a history of seizures or convulsions, excluding febrile convulsions in childhood
  * Subjects with underlying muscle disease or a history of muscle disease (for example, polymyositis or rhabdomyolysis)
  * Evidence or recent history of significant active psychiatric disease such as schizophrenia, depression, or bipolar disorder
  * Recent immobilization or major trauma to the legs within 6 months
  * Knee or hip replacement or lower extremity amputation
  * Participate in, or have participated within 3 months of study drug administration, a regular resistance training program or plan to participate in an exercise program during the study
  * Actively working in a physically demanding profession
  * Have contraindications for the Magnetic Resonance Imaging (MRI) scan
  * Tattoos on the right leg if the tattoos are at least 20 years old and may have iron-containing pigments
  * Electrocardiogram (ECG) considered outside the normal limits for the study population by the investigator and relevant for interpretation or indicating cardiac disease
  * Clinically significant abnormality in neurologic or neurocognitive examinations at screening

Ages: 24 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single IV Dose 70 mg LY2495655: Single 70 milligram (mg) dose LY2495655 administered intravenously (IV)
- Multiple SC Dose 140 mg LY2495655: 140 mg of LY2495655 administered subcutaneously (SC) every 2 weeks for 8 weeks (total 5 of doses)
- Multiple SC Dose 420 mg LY2495655: 420 mg dose of LY2495655 administered subcutaneously (SC) every 2 weeks for 8 weeks (total 5 of doses)
Period: Overall Study
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655 | Single IV Dose Placebo | Multiple SC Dose Placebo
Started | 6 | 9 | 10 | 10 | 2 | 10
Received at Least 1 Dose of Study Drug | 6 | 9 | 10 | 10 | 2 | 10
Completed | 6 | 9 | 9 | 9 | 2 | 9
Not Completed | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Sponsor decision | 0 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655 | Single IV Dose Placebo | Multiple SC Dose Placebo | Total
Number analyzed (Participants) | 6 | 9 | 10 | 10 | 2 | 10 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (4.2) | 64.6 (7.2) | 61.2 (6.9) | 60.3 (3.3) | 48.0 (11.3) | 65.0 (9.2) | 60.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 3 | 1 | 4 | 17
  Male | 4 | 6 | 6 | 7 | 1 | 6 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Japanese | 6 | 9 | 10 | 10 | 2 | 10 | 47
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 9 | 10 | 10 | 2 | 10 | 47
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 66.48 (8.55) | 62.04 (7.31) | 63.29 (12.56) | 64.05 (9.08) | 57.15 (12.66) | 62.90 (12.36) | 63.28 (10.05)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 167.83 (6.81) | 163.57 (4.97) | 162.01 (8.11) | 162.70 (6.20) | 165.65 (15.06) | 164.52 (6.57) | 163.89 (6.82)
International Physical Activity Questionnaire (IPAQ) [Mean (Standard Deviation); unit: MET-minutes per week] — IPAQ assessed physical activity, walking, moderate-intensity activities and vigorous-intensity activities. The total IPAQ score is computed by weighting each type of activity by its energy requirements defined in Metabolic Equivalent Tasks (METs). A MET-minute score is multiplied by an activity by the minutes performed (MET-minute=kilocalories for a 60 kilogram person). Data is expressed as MET-min per week: MET level x minutes of activity x events per week. A MET-min per week score below 600 is considered low physical activity (sedentary) and a score above 600 is high physical activity.
  MET-minutes per week | 1829.25 (1619.29) | 278.11 (341.65) | 130.80 (214.24) | 331.50 (301.53) | NA (NA) — Only 2 participants; 618 (min) and 693 (max); mean was not calculated due to it's a center of those values. | 108.40 (198.18) | 436.10 (803.71)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant effects are defined as treatment emergent adverse events (TEAEs) which in the opinion of the investigator are thought to be possibly related to study drug. A summary of serious and all other non-serious adverse events (whether or not related to study drug) is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion (up to 135 days)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655 | Single IV Dose Placebo | Multiple SC Dose Placebo
Number analyzed (Participants) | 6 | 9 | 10 | 10 | 2 | 10
Participants | 0 | 0 | 7 | 4 | 0 | 2

2. Secondary Outcome: Pharmacokinetics, Maximum Concentration (Cmax)
Time Frame: Single Dose:Day 1:Predose,10 minutes before end,2,6,12,24,48,192,360,528,696,1032,1368and2040 hours(hrs)Postdose;Multiple Dose:Day 1:Predose,24,48,96,168,264,360,528,696,1032hrs Postdose; Day57:Predose,24,48,96,168,336,672and1680hrs Postdose
Population: All participants who received study drug and had evaluable Cmax data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per milliliter (pmol/mL)
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655
Number analyzed (Participants) | 6 | 9 | 10 | 10
picomoles per milliliter (pmol/mL)
  Day 1 | 192 (7) | 8.11 (41) | 102 (80) | 303 (42)
  Day 57: number analyzed (Participants) | 0 | 9 | 9 | 9
  Day 57 |  | 23.8 (36) | 304 (32) | 1060 (24)

3. Secondary Outcome: Pharmacokinetics, Area Under the Concentration Versus Time Curve (AUC)
Description: Area under the concentration curve (AUC) time zero to infinity (0-inf) was calculated for single dose administration and AUCtau (AUCτ) at steady state was calculated for multiple dose administration.
Time Frame: as for outcome 2
Population: All participants who received study drug and had evaluable AUC data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour per milliliter(nmol*h/mL)
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655
Number analyzed (Participants) | 6 | 9 | 10 | 10
nanomoles*hour per milliliter(nmol*h/mL)
  Day 1 | 50.5 (11) | 2.32 (34) | 24.0 (59) | 79.8 (40)
  Day 57: number analyzed (Participants) | 0 | 9 | 9 | 9
  Day 57 |  | 6.82 (39) | 88.7 (32) | 319 (23)

4. Secondary Outcome: Pharmacokinetics, Time of Maximum Observed Drug Concentration (Tmax)
Time Frame: as for outcome 2
Population: All participants who received study drug and had evaluable Tmax data were analyzed.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655
Number analyzed (Participants) | 6 | 9 | 10 | 10
hours (h)
  Day 1 | 0.58 [0.50 to 2.50] | 168 [48 to 335] | 168 [96 to 264] | 167 [48 to 335]
  Day 57: number analyzed (Participants) | 0 | 9 | 9 | 9
  Day 57 |  | 48.0 [24.0 to 168] | 96.0 [47.8 to 168] | 96.0 [48.0 to 168]

5. Secondary Outcome: Percentage Change in Thigh Muscle Volume
Description: Thigh muscle volume was determined by Magnetic Resonance Imaging (MRI) scan of the right leg thigh muscle. Percentage change in thigh muscle volume=(time point value-baseline value)*100. Change from baseline for muscle volume was analyzed using mixed model repeated measures (MMRM) model with fixed effects of treatment, time and treatment*time interaction and a random effect of subject where baseline values were included as a covariate.
Time Frame: Baseline, Day 22 for a single dose arm/ baseline, Days 22 and 71 for multiple dose arms
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655 | Single IV Dose Placebo | Multiple SC Dose Placebo
Number analyzed (Participants) | 6 | 9 | 10 | 10 | 2 | 10
percentage change
  Day 22 | 0.30 (2.33) | 0.40 (1.40) | 1.51 (2.48) | 1.80 (1.46) | NA (NA) — Only 2 participants, thus not calculated | -1.15 (1.81)
  Day 71: number analyzed (Participants) | 0 | 9 | 9 | 9 | 0 | 9
  Day 71 |  | 1.33 (2.47) | 2.88 (2.39) | 3.48 (2.84) |  | -1.22 (2.97)

ADVERSE EVENTS:
Arm/Group | Single IV Dose 70 mg LY2495655 | Multiple SC Dose 17.5 mg LY2495655 | Multiple SC Dose 140 mg LY2495655 | Multiple SC Dose 420 mg LY2495655 | Single IV Dose Placebo | Multiple SC Dose Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/10 | 0/10 | 0/2 | 0/10
Other Adverse Events (participants affected / at risk) | 4/6 | 9/9 | 10/10 | 10/10 | 2/2 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single IV Dose 70 mg LY2495655 (N=6) | Multiple SC Dose 17.5 mg LY2495655 (N=9) | Multiple SC Dose 140 mg LY2495655 (N=10) | Multiple SC Dose 420 mg LY2495655 (N=10) | Single IV Dose Placebo (N=2) | Multiple SC Dose Placebo (N=10)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 2 (2) | 6 (8) | 3 (6) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 3 (7) | 2 (3) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 3 (3) | 5 (9) | 4 (4) | 3 (4) | 0 (0) | 3 (4)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Sleep phase rhythm disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days